CLINICAL TRIAL: NCT01284699
Title: Evaluation of the Safety and Efficacy of Bilateral Subthalamic Nucleus (SNT) Radiosurgery in Idiopathic Severe Parkinson's Disease Fulfilling Inclusion Criteria for STN Deep Brain Stimulation and Presenting With a Contraindication to Intracerebral Electrode Implantation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-A01227-50; 2009/34
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease; With Inclusion Criteria for STN Deep Brain Stimulation; Presenting a Contraindication to Intracerebral Electrode Implantati
Keywords: Parkinson; contraindication to Intracerebral electrode implantation; Gamma Knife radiosurgery
MeSH Terms: conditions — Parkinson Disease | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gamma Knife radiosurgery — For patients presenting a contraindications for anaesthesia or electrode implantation, operate their brain without opening the skull without infection or bleeding risk.

SUMMARY:
The goal of our trial is to evaluate the tolerance and efficacy of the STN radiosurgery in Parkinsonian patients presenting with the inclusion criteria for the STN stimulation but presenting also with clear contraindications to the implantation of the deep brain electrodes.

DETAILED DESCRIPTION:
Subthalamic nucleus (SNT) deep brain stimulation (DBS) is the reference treatment for severe drug resistant Parkinson's disease, responsible to dopaminergic therapy, to the state of complication. The efficacy of this therapeutic approach has transformed the functional prognosis of these patients. Unfortunately, those of the patients presenting with contraindications for anaesthesia or electrode implantation are excluded of these therapeutic hope.

Gamma Knife radiosurgery is a neurosurgical procedure going to operate in the brain of the patients without opening the skull without infection or bleeding risk.

Gamma Knife radiosurgical treatment will be done in two separate times (GK1 and GK2). Treatment of the second side (GK2) will be done at least 12 months after the treatment of the first side (GK1), in the same methodology as the first treatment. The major risk of onset of acute ballism although low is planned to be managed by the standard protocol by the recruiting team involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with contraindications for anaesthesia or electrode implantation

Exclusion Criteria:

* contraindications for a surgical treatment
* Pregnant or breast-feeding women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and efficacy | 48 months
  Feasibility of this step is mandatory on the organization of a true randomized comparative trial witch should bring a higher lever of evidence, but in the present state immature from ethical point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Jean -Marie REGIS, Professor, Principal Investigator — APHM
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France